CLINICAL TRIAL: NCT05299268
Title: The Influence of Pain on Exercise-Induced Hypoalgesia in Healthy Women
Brief Title: Influence of Pain on Exercise-induced Hypoalgesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aalborg University (Other)
Collaborators: University of Southern Denmark (Other)
Responsible Party: Principal Investigator, Steffan Wittrup Christensen, Associate Professor, Aalborg University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: S-20210184
Record Dates: First submitted 2022-02-25; First posted 2022-03-28 (Actual); Last update posted 2022-04-20 (Actual); Status verified 2022-04

CONDITIONS: Pain; Healthy
MeSH Terms: conditions — Pain | interventions — Saline Solution, Hypertonic; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: This study is a 2-arm randomized controlled cross-over trial with 1-7 days between arms
Who Masked: Participant, Investigator
Masking Description: Assessor and participants will be blinded to the order of injections.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pain (hypertonic saline) (Experimental): Injection (1 ml) of painful hypertonic saline (5.8%) prior to performance of the 1x3 min Seated Isometric Knee Extension
  Interventions: Behavioral: Pain (hypertonic saline)
- No pain (isotonic saline) (Placebo Comparator): Injection (1 ml) of non-painful isotonic saline (0.9%) prior to performance of the 1x3 min Seated Isometric Knee Extension
  Interventions: Behavioral: No pain (Isotonic saline)

INTERVENTIONS:
Behavioral: Pain (hypertonic saline) — A bolus injection (1 ml) of hypertonic saline (5.8%) is injected into the dominant vastus medialis muscle 20 cm proximal from the basis of patella before performance of the 1x3 min Seated Isometric Knee Extension.
  Arms: Pain (hypertonic saline)
Behavioral: No pain (Isotonic saline) — A bolus injection (1 ml) of isotonic saline (0.9%) is injected into the dominant vastus medialis muscle 20 cm proximal from the basis of patella before performance of the 1x3 min Seated Isometric Knee Extension
  Arms: No pain (isotonic saline)

SUMMARY:
The purpose of this study is to investigate how acute pain induced by hypertonic saline prior to exercise influence the magnitude of exercise-induced hypoalgesia after 1x3 min seated isometric knee extension exercise in healthy women. The study is a blinded randomized cross-over trial The results from the study may be of great importance to the understanding of exercise-induced hypoalgesia, and whether the presence of pain affects the effects of exercise.

DETAILED DESCRIPTION:
Exercise is recommended to promote and maintain health and as treatment for more than 25 chronic diseases and pain conditions.

The mechanisms underlying pain relief of exercise are largely unknown but may be related to the modulation of central descending pain inhibitory pathways after acute exercise bouts. Exercise-induced hypoalgesia (EIH) is typically assessed as the temporary change in pressure pain thresholds (PPT) after a short acute exercise bout and EIH is seen as a proxy of descending pain inhibitory control. In general, EIH seems hypoalgesic (functional) in asymptomatic subjects. A hyperalgesic (impaired) EIH response has been reported in different chronic pain populations, although a functional EIH response also has been reported in subgroups of knee osteoarthritis patients. This implies differences in the acute response to exercise between healthy (pain-free) subjects and chronic pain patients, but it is still unknown whether the presence of pain itself affects the pain alleviating response (i.e. the EIH response) to acute exercise.

It is hypothesized that acute pain will decrease the EIH response magnitude following hypertonic saline injection compared with the control injection. This study will increase the insight into the EIH mechanisms in healthy subjects in general, and how the presence of pain affects the body's own ability to modulate pain during exercise.

ELIGIBILITY:
Inclusion Criteria:

* Pain-free
* Understands and writes Danish

Exclusion Criteria:

* Pregnancy
* Previous addictive behaviour defined as abuse of hash, opioids or other euphoric substances.
* Previous painful or mental illnesses, neurological or circulatory diseases in the form of heart or lung disease.
* Surgery in the lower extremities within the last 12 months
* Chronic or actual pain on the days of testing
* Under the influence on the days of testing
* Inability to cooperate

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2022-03-08 (Actual); Primary Completion 2022-04-12 (Actual); Study Completion 2022-04-12 (Actual)

PRIMARY OUTCOMES:
Change in pressure pain threshold will be assessed over the dominant quadriceps muscle | Baseline, Day 2 (within 1 week of baseline), Day 3 (within 1 week of Day 2)
  Between group comparison of the primary outcome, which is change in pressure pain threshold over the dominant quadriceps muscle before and after performing seated isometric knee extension.
  Pressure pain threshold is measured with a handheld pressure algometer.

SECONDARY OUTCOMES:
Pressure pain threshold at the non-dominant quadriceps muscle and non-dominant trapezius muscle | Baseline, Day 2 (within 1 week of baseline), Day 3 (within 1 week of Day 2)
  Between group comparison of the secondary outcome, which is change in pressure pain threshold at the non-dominant quadriceps muscle and non-dominant trapezius muscle from before Seated Isometric Knee Extension to after Seated Isometric Knee Extension.
  Pressure pain threshold is measured with a handheld pressure algometer.
Pain Intensity in dominant thigh | Assessed before and immediately after hypertonic and isotonic saline injection as well as 1, 2 and 3 minutes into the Seated Isometric Knee Extension, and immediately after the end of the seated isometric knee extension
  Pain intensity is assessed with numerical rating scales with 0 = no pain and 10 = maximal pain.

OTHER OUTCOMES:
Pressure pain threshold at the dominant and non-dominant thigh as well as non-dominant trapezius muscle | Before and after determining maximal voluntary contraction on the fist test day and prior to saline injections
  Pressure pain threshold is measured with a handheld pressure algometer.
Rating of perceived exertion (RPE) | Assessed 1, 2 and 3 minutes into the Seated Isometric Knee Extension
  Perceived exertion is assessed with Borg RPE scale with 6 = no exertion and 20 = maximal exertion
Quantifying the individual´s pain experience | Baseline
  Quantifying the individual´s pain experience will be assessed using the Pain Catastrophizing Scale (PCS) at the first session. The pain catastrophizing scale have 13 sentences regarding pain-related thoughts. Participants are asked to indicate how well each sentence applies for them: 0 = not at all, 1 = to a slight degree, 2 = to a moderate degree, 3 = to a great degree and 4 = all the time. A higher score is worse
Pain experience | Day 3 (within 2-3 weeks of the initial session)
  Participants will be interviewed at the end of the study regarding the experience of pain during the study. The interview will be conducted after all other experimental procedures have been completed.

CONTACTS AND LOCATIONS:
Overall Officials: Steffan WM Christensen, PhD, Principal Investigator — Aalborg University
Locations (1):
- Dept. Of Health Science and Technology, Aalborg University, Aalborg, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mohrsen A, Lund H, Rasmussen SZ, Vaegter HB, Vela J, Hansen S, Christensen SWM. Acute exercise of painful muscles does not reduce the hypoalgesic response in young healthy women - a randomized crossover study. Scand J Pain. 2023 May 4;23(3):599-607. doi: 10.1515/sjpain-2022-0127. Print 2023 Jul 26. PMID 37137551